CLINICAL TRIAL: NCT01374126
Title: Azithromycin Combination Therapy for the Treatment of Severe Malaria - A Pilot Safety and Efficacy Study in Uncomplicated Falciparum Malaria in Bangladesh
Brief Title: Azithromycin Combination Therapy for the Treatment of Severe Malaria
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Collaborators: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Responsible Party: Principal Investigator, Harald Noedl, Assoc. Prof. Dr., Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PR-11019
Record Dates: First submitted 2011-06-10; First posted 2011-06-15 (Estimated); Last update posted 2013-08-23 (Estimated); Status verified 2013-08

CONDITIONS: Falciparum Malaria
MeSH Terms: conditions — Malaria, Falciparum | interventions — Artesunate; Azithromycin

ARMS (2):
- Azithromycin-Artesunate (Experimental)
  Interventions: Drug: Azithromycin + Artesunate
- Control (artesunate alone) (Active Comparator)
  Interventions: Drug: Artesunate

INTERVENTIONS:
Drug: Artesunate — Artesunate alone
  Arms: Control (artesunate alone)
Drug: Azithromycin + Artesunate — Combination of azithromycin + artesunate
  Arms: Azithromycin-Artesunate

SUMMARY:
A randomized controlled trial to assess the safety and efficacy of azithromycin combination therapy for use in severe malaria. This pilot trial will be conducted in uncomplicated malaria patients in southeastern Bangladesh.

ELIGIBILITY:
Inclusion Criteria:

Male and female participants with a diagnosis of acute falciparum malaria meeting all criteria listed below may be included in the study:

1. Acute symptomatic falciparum malaria infection with a parasite density of 100 to 100,000 asexual parasites/uL as determined on the screening smear with fever (defined as ≥37.5ºC), or reported history of fever within the last 48 hours.
2. Age: 8-65 years old
3. Males or females. All females over the age of 12 are required to have a negative human chorionic gonadotropin (hCG) pregnancy test (urine). All females of childbearing potential (not surgically sterile, or less than two years menopausal) are required to use an acceptable method of contraception, such as implant, injectable, oral contraceptive(s) with additional barrier contraception, intrauterine device, sexual abstinence, or vasectomized partner, throughout the study
4. Written informed consent obtained
5. Willing to stay under close medical supervision for the study duration
6. Otherwise healthy outpatients

Exclusion Criteria:

Participants presenting with any of the following will not be included in the study:

1. Pregnant women, nursing mothers, or women of childbearing potential who do not use an acceptable method of contraception (as described in Inclusion Criteria, #3)
2. Mixed malaria infection on admission by malaria smear
3. A previous history of intolerance or hypersensitivity to the study drugs artesunate, azithromycin or to drugs with similar chemical structures
4. Malaria drug therapy administered in the past 30 days by history
5. History of significant cardiovascular, liver or renal functional abnormality or any other clinically significant illness, which in the opinion of the investigator would place them at increased risk.
6. Symptoms of severe vomiting (no food or inability to take food during the previous 8 hours).
7. Signs or symptoms of severe malaria (as defined by WHO 2003)
8. Unable and/or unlikely to comprehend and/or follow the protocol

Ages: 8 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2011-07; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability (Number of Participants with Adverse Events) | 42 days
Adequate Clinical and Parasitological Response (ACPR) on Days 28 and 42 | 42 days

CONTACTS AND LOCATIONS:
Locations (1):
- MARIB, Bāndarban, Bangladesh